CLINICAL TRIAL: NCT05655884
Title: The Effect of Listening To Music And Foot Reflexology on Nausea, Pain And Anxiety in Children During Perioperative Period
Brief Title: The Effect of Listening To Music And Foot Reflexology in Children During Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilek Kucuk Alemdar, Associate Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK117
Record Dates: First submitted 2022-11-28; First posted 2022-12-19 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Period
Keywords: Perioperative Period; Pain; Children; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This research was planned as randomized controlled, experimental.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research will be structured according to the CONSORT 2010 checklist of information to include when reporting a randomised trial (Schulz et al., 2010) to facilitate clarity, integrity, and transparency. The assignment of children to groups will be made using the "simple randomization method". Children will not be informed about which group they are in (playing music, foot reflexology, control). The data collection tools of the study will be filled by the child, the parent, and an experienced university graduate nurse working in the day surgery clinic independent of the research. The nurse will be informed by the researcher about the scales to be used in the research. The researcher will not be involved in the data collection process, he will only observe the process. In addition, the database of the research will be created by a university graduate statistician working in a statistical center independent of the research, apart from the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Listening Application (Experimental): Children in this group; 15 minutes before going to the surgery, the child's favorite and chosen music piece will be loaded onto the mp3 player and played by the researcher (who has received music therapy training) via the "creatone music pillow" for 15 minutes.
  Interventions: Other: Music Listening Application
- Foot Reflexology Practice (Experimental): Children in this group; Before going to the surgery, foot reflexology will be applied by the researcher (who has received reflexology training), only to the left foot, for 10 minutes.
  Interventions: Other: Foot Reflexology Practice:
- Control Group (No Intervention): Children in this group will not be subjected to any non-pharmacological application to reduce nausea, pain and anxiety before and after surgery. They will receive routine perioperative care administered in the clinic.

INTERVENTIONS:
Other: Music Listening Application — 15 minutes before going to the surgery, the child's favorite and chosen music piece will be loaded onto the mp3 player and played by the researcher via the "creatone music pillow" for 15 minutes. After the child returns to the service from the recovery room (the room where the patient is observed in the operating room for a certain period of time until he recovers from the surgery and his general condition is stable), and after he regains consciousness, music will be played by the music group again for 15 minutes.
  Arms: Music Listening Application
Other: Foot Reflexology Practice: — Children in this group; Before going to the surgery, foot reflexology will be applied by the researcher, only to the left foot, for 10 minutes. After the child returns to the service from the recovery room (the room where the patient is observed in the operating room for a certain period of time until he recovers from the surgery and his general condition is stable), and after he regains consciousness, foot reflexology will be applied again, only on the left foot, for 10 minutes.
  Arms: Foot Reflexology Practice

SUMMARY:
The population of the research will be children between the ages of 7 and 12 who underwent day surgery at the Pediatric Surgery Clinic of the Gynecology and Childhood Hospital of Ordu University Training and Research Hospital. The sample of the study will consist of 99 children who have undergone a day surgery operation between the specified dates, who meet the case selection criteria and agree to participate in the study.

DETAILED DESCRIPTION:
First of all, the hospitalized children and their parents will be informed about the study. Verbal and written consent will be obtained from the child and his/her parents who agreed to participate in the study before starting the study. "Child and Parent Descriptive Information Form, Baxter Nausea Scale-BARF, Multidimensional Perioperative Anxiety Scale in Children and Children's Emotional Indicator Scale will be administered to all children in the experimental and control groups 30 minutes before the operation (1st measurement). Before going to the operation, the music listening group will listen to music with a music pillow for 15 minutes, foot reflexology will be applied for 10 minutes to the foot reflexology group, and no application will be made to the control group. 10 minutes after the application, Baxter Nausea Scale-BARF, Multidimensional Perioperative Anxiety Scale in Children and Children's Emotional Indicator Scale will be administered again to all three groups (experimental and control) (2nd measurement). When the child comes to the service from the recovery unit after the surgery and after the necessary medical intervention (60th minute postoperatively), all scales will be applied (3rd measurement) and then the music listening group will be listened to with a music pillow for 15 minutes, reflexology will be applied to the foot reflexology group for 10 minutes, and the control group will be no application will be made and after 10 minutes all the scales will be re-administered to the experimental and control groups (4th measurement). Finally, 30 minutes before the child is discharged. First, all scales will be applied to the experimental and control groups again and an evaluation will be made with these results (5th measurement).

ELIGIBILITY:
Inclusion Criteria:

* - The child is between 7-12 years old,
* The child is hospitalized for general anesthesia and surgical operation,
* Parents and children are willing to participate in the research,
* The integrity of the tissue in the foot of the child is intact,
* The child does not have visual, hearing and mental disabilities,
* Parents and children give written and verbal consent,

Exclusion Criteria:

* The child has a hearing problem,

  * The child's hemodynamics is unstable,
  * The child has eye surgery, orthopedic surgery, inner ear surgery, adenoidectomy, tonsillectomy,
  * The child and the parent do not understand and speak Turkish easily,
  * The child is not at the level of mental development to be able to answer the questions asked,
  * Development of a high-risk condition in the child in the postoperative period,
  * Absence of a primary caregiver,
  * The child has a history of analgesic or narcotic substance use within 24 hours before surgery.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Baxter Nausea Scale- BARF Score | Nausea and vomiting change in the perioperative period.
  A score of 0 from the scale indicates that there is no nausea- vomiting, and a score of 10 indicates that there is nausea-vomiting
Eastern Ontario Children's Hospital Pain Scale | Pain change in the perioperative period.
  The total score from the scale is evaluated as the lowest 4 points and the highest 13 points. A high total score from the scale indicates that the child has high postoperative pain
Multidimensional Perioperative Anxiety Scale (MCPSPS) | Anxiety change in the perioperative period.
  The scale is a visual analog scale consisting of 5 items and scored between 0-100, prepared for children
  aged 7-13 who will undergo day surgery. An increase in the score obtained from the scale indicates that the child's perioperative anxiety increases.
Children's Emotional Indicator Scale (CBRS) | Emotional change in the perioperative period.
  As the scores obtained from the scale increase, negative emotional indicators increase. The rating is between 5-25 points.

SECONDARY OUTCOMES:
Heart rate (HR) | Heart rate in the perioperative period.
  It was created to monitor the heart rate (HR) of children in the perioperative period.
body temperature | Body temperature change in the perioperative period.
  body temperature of children in the perioperative period.
oxygen saturation (SpO2) | SpO2 change in the perioperative period.
  oxygen saturation (SpO2) of children in the perioperative period.
blood pressure | Blood pressure change in the perioperative period.
  blood pressure of children in the perioperative period.
respiratory rate | respiratory rate change in the perioperative period.
  respiratory rate of children in the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK KÜÇÜK ALEMDAR, Study Director — Ordu University
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No